CLINICAL TRIAL: NCT06845514
Title: High Blood Pressure and Effect of Acute Resistance Training: Influence of Different Load Intensities on Postexercise Hypotension and Ambulatory Blood Pressure in Aging Females
Brief Title: Impact of Resistance Training Intensity on Blood Pressure
Acronym: HEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-5649
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure Management; Blood Pressure Monitoring, Ambulatory; Blood Pressure, High; Blood Pressure
Keywords: resistance training; ambulatory blood pressure; aging females; load intensity; perceived effort
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Each participant will perform 3 experimental conditions (control condition; low-load resistance exercise; high-load resistance exercise).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition LL-RE (Experimental): Low-load resistance exercise
  Interventions: Other: Condition LL-RE
- Condition HL-RE (Experimental): High-load resistance exercise
  Interventions: Other: Condition HL-RE
- Condition CON (Sham Comparator): Control condition
  Interventions: Other: Control

INTERVENTIONS:
Other: Condition LL-RE — LL-RE condition will consist of a 5-minute warm-up (slow-paced walking) and the following exercises: leg press, chest press, leg curl, and seated row. Three sets will be performed for each exercise with a 3-minute rest period between sets/exercises. Each exercise will be executed through a full range of motion, with participants encouraged to follow a 2-sec eccentric phase (guided by a mobile app metronome and supervised by an exercise physiologist) and to perform the concentric phase as fast as possible. Participants will be informed to: stop the set when they perceive to have reached the RIR target.
  • LL-RE: The low load intensity protocol consists of 3 sets of each exercise at 50% 1-RM, performed until reaching a hard perceived effort intensity (i.e., RIR-2).
  Arms: Condition LL-RE
Other: Control — Control condition: During the control condition, participants will sit quietly in a room maintained at a temperature of 22-24°C to prevent any influence on blood pressure values, for 60 minutes. During this period, they will perform a standardized non-fatiguing cognitive task: watching Earth, a documentary following the migration paths of four animal families.
  Arms: Condition CON
Other: Condition HL-RE — HL-RE condition will consist of a 5-minute warm-up (slow-paced walking) and the following exercises: leg press, chest press, leg curl, and seated row. Three sets will be performed for each exercise with a 3-minute rest period between sets/exercises. Each exercise will be executed through a full range of motion, with participants encouraged to follow a 2-sec eccentric phase (guided by a mobile app metronome and supervised by an exercise physiologist) and to perform the concentric phase as fast as possible. Participants will be informed to: stop the set when they perceive to have reached the RIR target.
  • HL-RE: The high load intensity protocol consists of 3 sets of each exercise at 80% of 1-RM, performed until reaching a hard perceived effort intensity (i.e., RIR-2).
  Arms: Condition HL-RE

SUMMARY:
The goal of the clinical trial is to understand the effect of two resistance training protocols employing different loading intensities (% of 1 repetition maximum; 1-RM), but with standardized effort intensity (2 repetitions in reserve; RIR) on post-exercise and ambulatory blood pressure in aging females.

The main questions it aims to answer are:

* to examine the acute effects of low (50% 1-RM) and high (80% 1-RM) load intensity resistance exercise with a standardized high effort intensity on post-exercise hypotension and ambulatory blood pressure responses in aging females;
* deepen the understanding of the mechanisms underlying acute reductions in blood pressure in response to resistance exercise performed at different load intensities. To this end, autonomic activity will be estimated alongside the measurement of central arterial compliance (i.e., carotid artery), and serum biomarkers of endothelial function;
* document the affective valence and enjoyment associated with low (50% 1-RM) and high (80% 1-RM) load intensity resistance exercise when performed at a high perceived effort.

Researchers will compare the effect of: 1) a low load (LL-RE) intensity protocol consisting of 3 sets of each exercise at 50% 1-RM, performed until reaching a hard perceived effort intensity (i.e., RIR-2); 2) high load (HL-RE) intensity protocol consisting of 3 sets of each exercise at 80% of 1-RM, performed until reaching a hard perceived effort intensity (i.e., RIR-2); 3) and a control condition (CON) consisting of a standardized non-fatiguing cognitive task.

Participants will participate in:

* A preliminary assessment visit;
* Two familiarization visits to validate the exercise prescriptions;
* Three experimental visits (CON, LL-RE, HL-RE).

DETAILED DESCRIPTION:
Significant inconsistencies in the literature have led to resistance exercise often being overlooked as a method for managing high blood pressure and hypertension. The method of prescribing resistance exercise, whether it is based on load intensity (i.e., % of one-repetition maximum [1-RM]), perceived effort intensity (i.e., using a perception scale), or a combination of both, likely contributes to these inconsistencies. However, for inactive older adults, a growing number of studies suggest that lifting low loads (< 60% 1-RM) with high effort intensity, close to or until momentary muscle failure, is a promising approach for various health outcomes. However, it remains to be determined if this approach is acceptable and effective for blood pressure control. Moreover, there is a growing body of evidence suggesting marked sex differences in the acute and chronic blood pressure responses to resistance exercise, with women potentially benefiting more from low load intensity. This is particularly important because it has been reported that postmenopausal women achieve less adequate blood pressure control than men. Researchers propose to explore the effects of low-intensity resistance exercise (50% 1-RM) performed with high perceived effort intensity on post-exercise hypotension, known for its association with the long-term benefits of resistance training, and ambulatory blood pressure in postmenopausal women. Given that high-intensity load resistance training (≥ 75-80% 1-RM) is currently suggested and associated with chronic reductions in resting systolic blood pressure, researchers will also test whether this potential difference remains at a high load intensity (80% 1-RM) with high perceived effort intensity. These hypotheses will be tested while exploring the mechanisms related to post-exercise hypotension, taking into account enjoyment and affective valence, two important factors related to long-term exercise adherence.

Objective #1 (Primary): Examine the acute effects of low-intensity (50% 1-RM) and high-intensity (80% 1-RM) resistance exercise with standardized effort intensity (2 repetitions in reserve; [RIR]) on post-exercise hypotension and ambulatory blood pressure responses in aging women with normal-high resting blood pressure or hypertension.

Objective #2 (Secondary): Deepen the understanding of the underlying mechanisms of acute blood pressure reductions in response to resistance exercise performed at different load intensities. To this end, autonomic activity will be estimated alongside the measurement of central arterial compliance and serum biomarkers of endothelial function.

Objective #3 (Secondary): Document the affective valence and pleasure associated with low-intensity (50% 1-RM) and high-intensity (80% 1-RM) resistance exercise performed at high perceived effort.

A randomized crossover study including three experimental conditions will be conducted: CON, LL-RE (50% 1-RM), and HL-RE (80% 1-RM). A total of 36 women will be recruited according to these inclusion criteria: aged 50 to 70 years, absence of menstruation for 12 consecutive months, normal-high resting blood pressure (120 ≤ Systolic ≤ 139 mmHg and 80 ≤ Diastolic ≤ 89 mmHg) or stage 1 hypertension (140 ≤ Systolic ≤ 159 mmHg or 90 < Diastolic ≤ 99 mmHg), physically inactive (< 150 minutes of structured aerobic physical activity per week), and not engaging in regular resistance exercise (≥ 2 sessions per week) for more than 3 months during the year. Exclusion criteria include: orthopedic limitations or other contraindications to resistance exercise, scheduled surgery during the study, unstable hypertension (≥ 160/100 mmHg), diagnosis of type 2 diabetes, cardiovascular event in the past 6 months or sequelae preventing exercise, and initiation of hormonal replacement therapy (< 4 months) known to affect blood pressure. Eligible participants will be invited to the research center for a preliminary visit, and the following variables will be collected: resting heart rate, resting blood pressure, fasting metabolic profile, body composition, socio-demographic data, medical history, physical activity habits (questionnaires), and 1-RM tests to estimate the load to be used during experimental conditions. In the following two weeks (maximum), a familiarization period will take place, consisting of 2 sessions to familiarize participants with the exercises and the concept of perceived effort during this type of training. The experimental period will then begin with ≥ 72 hours between the 3 visits. During each experimental condition, blood pressure and heart rate variability will be assessed before and after the training session at regular intervals (every 20 minutes for 60 minutes), and ambulatory over 24 hours (non-dominant arm, every 20 minutes during the day and every 30 minutes at night). Blood samples and ultrasound measurements of carotid arterial compliance will also be collected before, immediately after the experimental portion (exercise), and 60 minutes later. In the 12 hours preceding the experimental conditions, participants must refrain from consuming caffeine and alcohol and limit moderate to vigorous physical activity. In the 24 hours following the experimental conditions, muscle soreness, food intake, and physical activity level will be assessed.

This study will be the first to determine if there are differences in the acute blood pressure responses to different load intensities during resistance exercises with a standardized effort intensity, a key variable in the prescription of resistance exercises for various health outcomes. The results will directly contribute to the existing knowledge on the impact of resistance exercise on blood pressure control in females, while taking into account patient-reported outcomes (affective valence and pleasure). These perspectives can provide valuable guidance to researchers and policymakers when evaluating the feasibility of implementing such an approach in clinical practice. Consequently, the results will help update exercise recommendations for blood pressure management and offer insights into the potential mechanisms responsible for hypotension.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 70 years;
* absence of menstruation for 12 consecutive months;
* normal-high resting blood pressure (120 ≤ Systolic ≤ 139 mmHg and 80 ≤ Diastolic ≤ 89 mmHg) or stage 1 hypertension (140 ≤ Systolic ≤ 159 mmHg or 90 < Diastolic ≤ 99 mmHg);
* physically inactive (< 150 minutes of structured aerobic physical activity per week);
* and not engaging in regular resistance exercise (≥ 2 sessions per week) for more than 3 months during the year.

Exclusion Criteria:

* orthopedic limitations or other contraindications to resistance exercise;
* scheduled surgery during the study;
* unstable hypertension (≥ 160/100 mmHg);
* diagnosis of type 2 diabetes;
* cardiovascular event in the past 6 months or sequelae preventing exercise;
* and initiation of hormonal replacement therapy (< 4 months) known to affect blood pressure.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In the case of initiation of a gender-affirming therapy known to influence blood pressure.
Enrollment: 36 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure post-exercise | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), each 20 min for 1 hour post-condition (t = 80, 100, 120 minutes)
  Oscillometric blood pressure monitor
Change in ambulatory blood pressure | During 24 hours after the condition
  Ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Heart rate variability | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), each 20 min for 1 hour post-condition (t = 80, 100, 120 minutes), during 24 hours after the condition
  Heart rate monitor
Carotid artery diameter as assessed by Cardiovascular Suite v4.6.1 | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Doppler ultrasound
Carotid artery distensibility as assessed by Cardiovascular Suite v4.6.1 | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Doppler ultrasound
Carotid artery blood flow velocity | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Doppler ultrasound
Serum endothelin-1 | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Enzyme-Linked Immunosorbent Assay
Serum endothelial nitric oxide synthase | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Enzyme-Linked Immunosorbent Assay
Serum catecholamines | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Enzyme-Linked Immunosorbent Assay
Salivary cortisol | Before the start of the condition (t = 0 minute), at the end of the condition (t = 60 minutes), 1 hour post-condition (t = 120 minutes)
  Enzyme-Linked Immunosorbent Assay
Affective valence | Before the start of the condition (t = 0 minute), during the condition (t = 30 minutes), at the end of the condition (t = 60 minutes)
  Valence Scale (-5, +5). Higher values are related to higher affective valence.
Enjoyment | At the end of the condition (t = 60 minutes)
  Physical Activity Enjoyment Scale (16, 80 points). Higher values are related to higher enjoyment.

OTHER OUTCOMES:
Velocity loss in concentric contraction speed | Continuously during the condition (t = 0 minute to t = 60 minutes)
  Video camera
Hematocrit/hemoglobin concentration | At the end of the condition (t = 60 minutes)
  Hemoglobin analyzer
Estimated daily energy expenditure | During 24 hours after the condition
  Accelerometer
Time spent in the different sedentary behaviors | During 24 hours after the condition
  Accelerometer
Food intake | In the 12 hours before the condition and during 24 hours after the condition
  Self-reported dietary logbook
Sleep quality | During 24 hours after the condition
  Likert scale (0, 7). Higher values are related to worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Eléonor Riesco, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No